CLINICAL TRIAL: NCT03720626
Title: Managed Access Program (MAP) Cohort Treatment Plan CSEG101A2001M to Provide Access to Crizanlizumab for Sickle Cell Disease Patients With History of Vaso-occlusive Crisis
Brief Title: MAP to Provide Access to Crizanlizumab, for Sickle Cell Disease Patients
Status: Available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CSEG101A2001M
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Sickle Cell Disease
Keywords: Sickle cell disease; sickle cell anemia; vaso-occlusive crisis; P-selectin; SEG101; crizanlizumab; monoclonal antibody; Anemia, Sickle Cell; HbS Disease; Hemoglobin SC Disease; Sickle Cell Disorders; Sickling Disorder Due to Hemoglobin S; Adult; Hb SS; Hb SC; Hb Sβ+-thalassemia; Hb Sβ0-thalassemia; Expanded Access Use; Pain Crisis; Compassionate Use
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises; Hemoglobin SC Disease | interventions — crizanlizumab

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: crizanlizumab — IV formulation with 30 min infusion, 5mg/kg dosage
  Other Names: SEG101

SUMMARY:
The purpose of this Cohort Treatment Plan is to allow access to crizanlizumab (SEG101) for eligible patients diagnosed with sickle cell disease (SCD) to prevent or reduce the frequency of vaso-occlusive crises (VOC). The patient's Treating Physician should follow the suggested treatment guidelines and comply with all local health authority regulations.

ELIGIBILITY:
Inclusion criteria

Written patient informed consent must be obtained prior to start of treatment, including all necessary consents (or their legal representatives, where applicable).

1. 1. Male or female, 12 years of age (inclusive) or older on the day of informed consent signature.
2. Confirmed diagnosis of sickle cell disease by hemoglobin electrophoresis or high performance liquid chromatography (HPLC) [performed locally]. All sickle cell disease genotypes are eligible (HbSS, HbSβ0, HbSC, HbSβ+, and others).
3. History of recurrent VOC as assessed by the Treating Physician.
4. Patients receiving HU/HC, L-glutamine (Endari), or other therapies as prevention therapy and continue to experience VOC while on any of these treatments.

   • Patients can continue taking the preventive therapy.
5. Patient is not a candidate to be treated with alternative treatment options or has discontinued alternative treatments due to unacceptable benefit risk as documented by the Treating Physician.
6. Patient must meet the following laboratory values prior to treatment:

   * Absolute Neutrophil Count ≥1.0 x 10^9/L
   * Platelets ≥ 75 x 10^9/L
   * Hemoglobin (Hgb) ≥ 4.0 g/dL
   * Estimated glomerular filtration rate ≥ 45 mL/min/1.73 m2 using CKD-EPI formula
   * Direct (conjugated) bilirubin ≤ 2.0 x ULN
   * Alanine transaminase (ALT) ≤ 3.0 x ULN
7. Received standard age-appropriate care for SCD, including an up-to-date record of immunizations, as per local requirements
8. Patients who are clinically stable and are in a non-crisis state at the time of treatment start

Exclusion criteria

Patients eligible for this Treatment Plan must not meet any of the following criteria:

1. Contraindication or hypersensitivity to any drug or metabolites from similar class as crizanlizumab drug or to any excipients of the drug formulation.
2. History of severe hypersensitivity reaction to other monoclonal antibodies, which in the opinion of the Treating Physician may pose an increased risk of serious infusion reaction.
3. Has documented immunogenicity to a prior biologic.
4. Pregnant or nursing women
5. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 15 weeks after stopping treatment. Highly effective contraception methods include:

   * Total abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
   * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before taking crizanlizumab. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
   * Male sterilization (at least 6 months prior to treatment). The vasectomized male partner should be the sole partner for that patient
   * Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
   * In case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before starting treatment.
   * Women of child bearing potential must be informed that taking the study treatment may involve unknown risks to the fetus if pregnancy were to occur during the study and agree that in order to participate in the MAP they must adhere to the contraception requirement for the duration of treatment.
6. Patients with bleeding disorders
7. Known history of testing positive for Human Immunodeficiency Virus (HIV) infection
8. Patients with active Hepatitis B infections (HBsAg positive)

   - Note: Patients with antecedent but no active Hepatitis B (i.e. anti-HBc positive, HBsAg and HBV-DNA negative) are eligible
9. Patients with positive test for hepatitis C ribonucleic acid (HCV RNA)

   - Note: Patients in whom HCV infection resolved spontaneously (positive HCV antibodies without detectable HCV-RNA) or those that achieved a sustained virological response after antiviral treatment and show absence of detectable HCV RNA ≥ 6 months (with the use of IFN-free regimes) or ≥ 12 months (with the use of IFN-based regimes) after cessation of antiviral treatment are eligible
10. Significant active infection or immune deficiency (including chronic use of immunosuppressive drugs)
11. Malignant disease. Exceptions to this exclusion include the following: malignancies that were treated curatively and have not recurred within 2 years prior to treatment; completely resected basal cell and squamous cell skin cancers and any completely resected carcinoma in situ
12. Has a serious mental or physical illness, which, in the opinion of the Treating Physician would compromise compliance to treatment.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

REFERENCES:
- [Derived] DeBonnett L, Joshi V, Silva-Pinto AC, Colombatti R, Pasanisi A, Arcioni F, Cancado RD, Sarp S, Sarkar R, Soliman W. Real-World Evidence of Crizanlizumab Showing Reductions in Vaso-Occlusive Crises and Opioid Usage in Sickle Cell Disease. Eur J Haematol. 2025 Feb;114(2):293-302. doi: 10.1111/ejh.14323. Epub 2024 Oct 29. PMID 39473076